CLINICAL TRIAL: NCT04597320
Title: The Effects of Esketamine Sedation Compared With Fentanyl Sedation in Pediatric Dental Patients: A Double Blind, Randomized Controlled Trial
Brief Title: Esketamine Sedation and Fentanyl Sedation in Pediatric Dental Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Yang Xudong, Chief of Department of Anesthesiology, Peking University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PKUSSIRB-202056103
Record Dates: First submitted 2020-09-10; First posted 2020-10-22 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Ketamine; Fentanyl; Sedation Complication
Keywords: Esketamine; Fentanyl; sedation; Pediatric dental patients
MeSH Terms: interventions — Fentanyl; Esketamine; Midazolam

STUDY DESIGN:
Intervention Model Description: Fentanyl group and Esketamine group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fentanyl group (Active Comparator): The fentanyl group was prepared by 1ug/kg fentanyl in 5ml normal saline, assembled with 5ml injection, labeled as "Anesthesia inducer". Midazolam 0.05mg/kg+ "Anesthesia inducer" was applied to all patients for procedural induction by intravenous injection. According to the MOAA/S score of the patients, midazolam could be added 0.5mg per time at more than 2 minutes until the MOAA/S score reached 3, the maximum infusion dose of midazolam was less than 10mg and less than 0.1mg/kg.
  Interventions: Drug: Fentanyl; Drug: Midazolam
- Esketamine group (Experimental): The esketamine group was prepared by 0.5mg/kg esketamine in 5ml normal saline, assembled with 5ml injection, labeled as "Anesthesia inducer". Midazolam 0.05mg/kg+ "Anesthesia inducer" was applied to all patients for procedural induction by intravenous injection. According to the MOAA/S score of the patients, midazolam could be added 0.5mg per time at more than 2 minutes until the MOAA/S score reached 3, the maximum infusion dose of midazolam was less than 10mg and less than 0.1mg/kg.
  Interventions: Drug: Esketamine; Drug: Midazolam

INTERVENTIONS:
Drug: Fentanyl — The fentanyl group was prepared by 1ug/kg fentanyl in 5ml normal saline, assembled with 5ml injection, labeled as "Anesthesia inducer".
  Arms: Fentanyl group
Drug: Esketamine — The esketamine group was prepared by 0.5mg/kg esketamine in 5ml normal saline, assembled with 5ml injection, labeled as "Anesthesia inducer".
  Arms: Esketamine group
Drug: Midazolam — Midazolam 0.05mg/kg+ "Anesthesia inducer" was applied to all patients for procedural induction by intravenous injection. According to the MOAA/S score of the patients, midazolam could be added 0.5mg per time at more than 2 minutes until the MOAA/S score reached 3, the maximum infusion dose of midazolam was less than 10mg and less than 0.1mg/kg.

SUMMARY:
Since the 1970s, ketamine has been used in clinical anesthesia treatment. Compared with ketamine, esketamine has a higher clearance rate, so it has a shorter recovery time after anesthesia. This feature also makes ketamine more suitable for pediatric dental patients.The purpose of this study was to investigate and compare the efficacy of esketamine sedation and fentanyl sedation in pediatric dental patients

ELIGIBILITY:
Inclusion Criteria:

* Age 6-14 years old.

  * Oral out-patient sedative treatment in our hospital.

    * BMI between 18 to 30 kg/m2. ④. ASA: I-II degree. ⑤. Sign the informed consent.

Exclusion Criteria:

* Patients who are allergic to esketamine, opioids, propofol, or have contraindications for these drug use.

  * Patients with mental illness or who are unable to cooperate.

    * Patients who have abnormal reaction to midazolam. ④. Patients who suffer from Apnea. ⑤. Patients who refuse to sign informed consent. ⑥. Patients who participated in other clinical trials within 4 weeks.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-12 (Actual)

PRIMARY OUTCOMES:
Hypoxemia | Day 0
  The incidence of intraoperative hypoxemia (Spo2<92%)
Midazolam use | Day 0
  The total use of midazolam

SECONDARY OUTCOMES:
Successful sedation | Day 0
  Success rate of sedation
Respiratory depression | Day 0
  Incidence of intraoperative respiratory depression and the need for airway support such as mandibular dragging
Agitation and delirium | Day 0
  The incidence of agitation and delirium during and after operation
Circulatory fluctuation | Day 0
  Occurrence of hypertension, hypotension, bradycardia, tachycardia and other side effects
Propofol requiring | Day 0
  Incidence of sedation requiring propofol
Time of successful sedation | Day 0
  The time when the MOAA/S score was equal to 3 points for the first time after patients were given anesthetic inducer
MOAA/S score in recovery room | Day 0
  MOAA/S score of patients every 15 minutes after entering the recovery room
The time for Modified Observer Assessment of Sedation Score(MOAA/S)>4 | Day 0
  The time for MOAA/S score to be greater than 4 since the end of clinical operation and the cessation of anesthetic infusion. MOAA/S is from 0 to 5, the higher of the score means the less sedative condition.
Directional force recovery time | Day 0
  Recovery time of directional force
Recall of intraoperative events | Day 0
  The child's recall of intraoperative events
Treatment comfort score | Day 0
  Patients' satisfaction score of treatment comfort. This score is from 0 to 10, the higher of the score means the more comfortable of the treatment patients received.
The incidence of complications | Day 1
  The incidence of patients suffered from pain, drowsiness, vomiting, nausea, mental emotion,within 1 day after treatment
Visual Analogue Scale(VAS) of pain in recovery room | Day 0
  Evaluate patients' VAS of pain every 15 minutes after entering the recovery room. This scale is from 0 to 10, the higher of the scale means the more painful patients feel.

CONTACTS AND LOCATIONS:
Overall Officials: Xudong Yang, MD, Study Chair — Department of anesthesiology of peking university school of stomatology
Locations (1):
- Peking University Hospital of Stomatology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code